CLINICAL TRIAL: NCT00718432
Title: Interventional Study of Geriatric Frailty, Osteoporosis, and Depression in a Community Based Randomized Trial.
Brief Title: An Interventional Study of Geriatric Frailty, Osteoporosis, and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: EC0970301
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Frailty; Osteoporosis; Depression
Keywords: Frailty; Osteoporosis; Depression
MeSH Terms: conditions — Frailty; Osteoporosis; Depression | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- UC group (Active Comparator): Usual care with education
  Interventions: Behavioral: Usual care with education
- ENIC group (IC group in 2009 study) (Experimental): Exercise and nutritional integrated care
  Interventions: Behavioral: Exercise and nutritional integrated care
- PSTIC group (IC group in 2009 study) (Experimental): Problem solving therapy integrated care
  Interventions: Behavioral: Problem solving therapy (PST) integrated care

INTERVENTIONS:
Behavioral: Exercise and nutritional integrated care — Besides the information sharing and the educational booklets, the ENIC group subjects are invited to take a structured exercise course at the participating hospital 3 times a week for 3 months. (twice a week for 24 weeks in 2009 study) The exercise program included warm up; a range of motion, stretching, and postural-correction activities; aerobic strengthening; balance; and cool down. The research team also inquired about the subjects' dietary compliance and responded to their dietary questions during the exercise sessions.
  Arms: ENIC group (IC group in 2009 study)
Behavioral: Usual care with education — The study educational booklet (plus CD-ROM in 2009 study) on frailty, depression, osteoporosis, healthy diets, exercise protocols, and coping strategies are given to the participants. UC group subjects will receive a 2-hour education based on the content of study booklet including 1-hour demonstration of study exercise program in 2009 study. Subjects are contacted monthly (bimonthly in 2009 study ) for frequencies of reading this booklet and the compliance on the suggested diet and exercise protocols. Subjects are also encouraged to follow with their primary care physicians for abnormal results identified from our assessments.
  Arms: UC group
Behavioral: Problem solving therapy (PST) integrated care — Besides the information sharing and the educational booklets, the PSTIC group subjects will receive 6 sessions of PST (within 12 weeks in pilot study, within 24 weeks in 2009 study) aiming at solving the 'here-and-now' problems contributing to their mood-related condition and helps increase their self-efficacy. If major depressions are found, subjects are referred to their primary care physicians for further medical managements.
  Arms: PSTIC group (IC group in 2009 study)

SUMMARY:
Frailty, osteoporosis, and depression are three highly prevalent geriatric syndromes. Having these conditions are associated with adverse outcome in physical health, mental health, quality of life, and daily functioning. They are associated with higher mortality rates as well as increased health care cost. Risk factors, pathogenesis, clinical phenotypes, and interventions of these three geriatric syndromes are often related. Frailty is often defined as accumulations of multi-system deficiencies with increased vulnerability to multiple worse outcomes. Multifactorial, interdisciplinary integrated care models targeting frail older adults may have positive impacts on measurements associated with not only frailty, but also depression, or osteoporosis. The objective of this proposed study is to conduct a randomized control trial (RCT) to exam the effectiveness of integrated interventions on multiple outcomes among community-dwelling Taiwanese elders with high risks for frailty and/or osteoporosis, depression. We also plan to determine the differential effects of intervention between urban and rural area.

DETAILED DESCRIPTION:
This is a three-year study. In the first year, we conducted a pilot study to test the feasibility of implementing integrated model on frailty, osteoporosis, depression, and other outcomes. Another objective is to determine optimal sample size for next level intervention in year 2 and 3 (2009 study).

Subjects are community-dwelling Taiwanese elders (65-79 years of age) living in Toufen Town in Miaoli County, Taiwan. Subjects are first screened with telephone interviews with the Chinese Canadian Study of Health and Aging _Clinical Frailty Scale (CCSHA_CFS). Eligible subjects are invited to a community hospital to be screened with the Health Study Phenotypic Classification of Frailty (CHS_PCF). Subjects scored ≥ 1 on the CHS_PCF are enrolled. With a 2 by 2 factorial design, subjects are first randomized into exercise/nutrition integrated care (ENIC) group and usual care (UC) group with education. Within each group, subjects are further randomized into problem solving therapy (PST) and usual care (UC) group with education by study care managers with pre-specified protocol. UC group subject received a study educational booklet with telephone follow up on compliance of booklet reading and suggested diet and exercise programs. Besides the booklets, ENIC group subjects received structured exercise 3 times/week with nutrition consultation as needed at hospital for 3 months while PST group subjects received 6 sessions of PST at hospital in 3 months.

Subjects were followed at 3, 6 and 12 months. Primary outcome is improvement of the CHS_PCF by at least one category (from pre-frail to robust, or from frail to pre-frail or robust) from baseline analysis. Secondary outcomes include the physical function and performance, cognition, depression, quality of life, healthcare resource utilizations and bone-mineral density (BMD). Intention-to-treat analysis was applied.

The pilot study enrolled 117 subjects, after analysis of the preliminary results, the study protocol for the second and third year (2009 study) is modified as follows:

1. The study is conducted at one urban (Wanhua) and one rural (Toufen) site with roughly 150 participants at each site.
2. Convenient samples referred from participant physicians' clinics instead of the population based samples in year 1 are used to decrease administration cost.
3. Telephone based first stage screening instrument will be modified and validated for face to face interview.
4. Longer intervention period (6-months) than year 1.
5. Interventions provided in ENIC and PSTIC groups are combined into a single integrated care (IC) group. Interventions for IC group and UC group are minor changed, as described below.

UC group: Inform the subjects about results of frailty, osteoporosis or depression assessment. The study educational booklet and CD-ROM on frailty, depression, osteoporosis, healthy diets, exercise protocols, and self-coping strategies will be given to participants. One 2-hour educational session is provided to participants to go through the booklet with demonstration of study exercise protocol. Subjects are encouraged to have balanced nutrition and regular exercises at home following the study protocol. Subjects were contacted bimonthly to check on how much they had read and watched the study material, and how well they had complied with the suggested diet and exercise protocols. However, it is at the subjects' discretion to discuss with their primary care physicians regarding the clinical interventions.

IC group: Subjects will receive all interventions provided to the UC group. Furthermore, subjects will take exercise/rehabilitation courses at the participating hospitals twice a week for 24 weeks and 6 sessions of problem solving treatment (PST). If subjects do not improve on any of the 5 indicators from the (CHSPCF), comprehensive geriatric assessments (CGAs) are applied to identify more potential modifiable factors for frailty for individualized managements.

Actual number of subjects enrolled in pilot study and 2009 study are 117 and 289 respectively and the total number of subjects enrolled in pilot study and 2009 study is 406.

ELIGIBILITY:
Inclusion Criteria:

* Scored 3-6 with the "Canadian Study of Health and Aging Clinical Frailty Scale (CSHA- CFS) Chinese Telephone Interview Version" (Telephone Interview Version is replaced by In-Person Interview Version in 2009 study)
* Frailty index ≥ 1

Exclusion criteria:

* Nursing home residents
* Cannot speak any of the following three dialogues: Mandarin, Taiwanese and Haga
* Hearing impairment interfering with communication or daily activities
* Visual impairment interfering with communication or daily activities.
* Cannot complete the screening instrument with the CSHA-CFS Chinese Telephone/In-Person Interview Version
* Scored 1, 2, or 7 with the CSHA-CFS Chinese Telephone/In-Person Interview Version
* Cognitive impairment defined as 3-item recall ≤ 1
* Functional Impairment defined as not able to walk for 5 meters without assistance
* Suicidal Ideation defined as Suicide Subscale of The Mini-International Neuropsychiatric Interview (M.I.N.I.) ≥ 6
* Alcohol abuse disorders active within the last year. (score ≥ 2 on the CAGE)
* Organic mental disorders (Seizure, brain tumor, brain surgeries), History of schizophrenia or bipolar diagnosed from psychiatrist

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 406 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
improvement of frailty | baseline, 3, 6, and 12 months
  Improvement of Cardiovascular Health Study Phenotypical Classification of Frailty (CHS_PCF) by at least one category (from pre-frail to robust, or from frail to pre-frail or robust) from baseline assessments.

SECONDARY OUTCOMES:
Bone Mineral Density | baseline and 12 months
  Dual-emission X-ray absorptiometry (DXA) of both Hip and spine
quality of life assessment | pilot study: baseline, 3, 6, and 12 months, 2009 study: baseline, 6, and 12 months
  EQ-5D index-Taiwan utility
QUALEFFO_31 | pilot study: baseline, 3, 6, and 12 months, 2009 study: baseline, 6, and 12 months
  pain, physical function,mental function
barthel index | pilot study: baseline, 3, 6, and 12 months, 2009 study: baseline and 12 months
PRIME-MD (only measured in pilot study) | baseline, 3, 6, and 12 months
  The Primary Care Evaluation of Mental Disorders
BDI-II (only measured in 2009 study) | baseline, 6, and 12 months
  Beck Depression Inventory Second Edition
health-resource utilization | pilot study: baseline, 3, 6, and 12 months, 2009 study: baseline, 6, and 12 months
Original Frailty Indicators | baseline, 3, 6, and 12 months
  Weight loss, Exhaustion, Low level physical activity, Slow walking speed, Weak grip strength
timed up and go | baseline, 3, 6, and 12 months
one leg stand time | baseline, 3, 6, and 12 months
dominant hand grip strength | baseline, 3, 6, and 12 months
dominant knee extension power | baseline, 3, 6, and 12 months
vitamin B12 in blood | pilot study: baseline and 12 month, 2009 study: baseline and 6 months
vitamin D in blood | pilot study: baseline and 12 month, 2009 study: baseline and 6 months
CRP in blood | pilot study: baseline and 12 month, 2009 study: baseline and 6 months
testosterone in blood | pilot study: baseline and 12 month, 2009 study: baseline and 6 months
IL-6 in blood | pilot study: baseline and 12 month, 2009 study: baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ken N Kuo, M.D., Study Chair — Natoinal Health Research Institutes; Ching-Yu Chen, M.D., Principal Investigator — Natoinal Health Research Institutes; Rong-Sen Yang, M.D., Principal Investigator — Natoinal Health Research Institutes; Keh-Ming Lin, M.D., Principal Investigator — Natoinal Health Research Institutes; Chao Agnes Hsiung, M.D., Principal Investigator — Natoinal Health Research Institutes
Locations (1):
- National Health Research Institutes, Zhunan, Taiwan

REFERENCES:
- [Derived] Chan DC, Tsou HH, Yang RS, Tsauo JY, Chen CY, Hsiung CA, Kuo KN. A pilot randomized controlled trial to improve geriatric frailty. BMC Geriatr. 2012 Sep 25;12:58. doi: 10.1186/1471-2318-12-58. PMID 23009149